CLINICAL TRIAL: NCT04269382
Title: Prospective, Multi-center Evaluation of the Accuracy of Non-invasive Measurement of Blood Pressure Using an Arm, Calf and Finger Cuff.
Brief Title: Accuracy of Non-Invasive Blood Pressure Measurements at the Arm, Calf , and Finger
Acronym: PANIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO 2019-09
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Hypotension and Shock; Hypertension; Intensive Care Unit
Keywords: Blood Pressure Determination
MeSH Terms: conditions — Hypotension; Shock; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined non-invasive and invasive BP measurements (Other): Patients will all undergo measurement of BP through 3 different techniques over a 30-min period: continuous noninvasive BP measurement (with the finger cuff and Clearsight™ device), repeated intermittent oscillometric NIBP measurements with a cuff placed around a calf or an arm, and continuous invasive BP measurement (through an indwelling arterial catheter).
  Interventions: Device: Combined non-invasive intermittent (oscillometric arm cuff), non-invasive continuous (finger cuff and ClearSight device), and invasive continuous (intra-arterial catheter) BP measurements

INTERVENTIONS:
Device: Combined non-invasive intermittent (oscillometric arm cuff), non-invasive continuous (finger cuff and ClearSight device), and invasive continuous (intra-arterial catheter) BP measurements — Continuous (finger cuff) noninvasive and invasive BP measurements, over a 30-min period. Pairs of noninvasive/invasive BP recorded each minute). In the same time, 3 pairs of oscillometric NIBP (cuff placed around a calf), and invasive BP measurements, at 30-sec intervals. The cuff is then placed around an arm and triplets of BP (arm cuff, finger cuff, intra-arterial catheter) will be taken over a 20-min period, at 3-min intervals and every time the invasive and/or the continuous finger cuff measurements cross the threshold of 65 mmHg for the mean BP. If clinically indicated, a cardiovascular intervention that can be either vascular volume expansion or initiation of vasoactive drug therapy, can be administered during this period. Finally, the cuff placed around the arm will be once again placed around the calf to take 3 pairs of oscillometric NIBP measurement with cuff placed around a calf, and simultaneous invasive BP measurement, at 30-second intervals.

SUMMARY:
The present study was designed to assess, in a population of patients admitted to the intensive care unit and already carrying an indwelling arterial catheter, the ability of combined continuous (ClearSight™) and intermittent (automatic cuff) non-invasive monitoring to detect low mean BP (<65mmHg). The intra-arterial measurement will be the reference measurement. As secondary objectives, the investigators will assess the ability of combined continuous (ClearSight™) and intermittent (automatic cuff) non-invasive monitoring to detect stage 2 hypertension, and to detect changes in BP during a cardiovascular intervention (as clinically indicated but not imposed by the study protocol). Additionally, the accuracy of both devices against the current international standard (ISO standard) will be assessed.

DETAILED DESCRIPTION:
The measurement of arterial blood pressure (BP) is of paramount importance when caring for critically ill patients, as BP, especially mean BP, is the driving force of blood flow through all the organs. The reference method is the invasive method that measures BP continuously and directly in an artery (most often the radial artery), through an indwelling arterial catheter. A popular, less invasive method, most often used in emergency situations or during the first hours of care in the intensive care unit (ICU), is the non-invasive oscillometric method (NIBP) using an arm cuff (some have shown that the cuff could also be placed around the calf, just above the ankle), that provides only intermittent measurements. In between the above 2 techniques, the place of continuous non-invasive BP monitoring devices using a different technology (plethysmography and volume clamp technique) and a cuff placed around a finger is uncertain. It would be interesting to evaluate whether the 2 non-invasive techniques (using arm or finger cuff) can be advantageously combined either to replace invasive monitoring or to reinforce non-invasive monitoring (in patients in whom an arterial catheter is not envisaged). In the critically ill patient, reliable detection of low BP is often the most important task assigned to BP monitoring devices, at least in the initial phase of management. It is conceivable that if the finger cuff (ClearSight™ device) was not infallible in measuring BP, low BP could still be detected sufficiently reliably by the finger cuff (even with weak accuracy), giving an early warning. The arm measurement could then confirm hypotension in a robust, on-demand manner, since the ability of the arm cuff to detect hypotension has already been demonstrated. The ability to detect hypotension using a combined non-invasive approach (finger and arm cuff) has never been explored with the ClearSight™ device. This combined approach could similarly detect high blood pressure or a rapid change in BP as a result of cardiovascular intervention. In addition, the automatic cuff cannot always be placed around the arm (presence of wounds, burns, fractures or surgery of the upper limb, venous catheter, etc.) for intermittent NIBP measurements, and is then placed around the calf. However, this commonly observed practice exposes the NIBP measurement to less accuracy. The finger cuff could be an alternative to the calf cuff. However, the accuracy of finger measurement has never been compared to the accuracy of oscillometric measurement at the calf.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised in one of the three recruiting intensive care units
* Patient already carrying an indwelling arterial catheter
* Stable BP over a 5-min period: no variation of mean BP above 10% and no change in vasopressor therapy

Exclusion Criteria:

* Brachial circumference > 42 cm.
* Any local fracture, wound, ischemic injury, infection, amputation, thrombophlebitis, that could prevent inflating a cuff around the arm or a finger
* Need of emergency therapy not compatible with the BP measurements schedule
* Asymmetry of mean BP between right and left arm (> 5 mmHg)
* Pregnancy
* Age < 18 years
* Patient under curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Discriminative power of the combined BP measurements with finger cuff and arm cuff to detect intra-arterial mean BP below 65 mmHg | 30 minutes
  Area under the receiver operating characteristics curve of the combined BP measurements with finger cuff and arm cuff to detect intra-arterial mean BP below 65 mmHg

SECONDARY OUTCOMES:
Discriminative power of the combined BP measurements with finger cuff and arm cuff to detect intra-arterial systolic hypertension | 30 minutes
  Area under the receiver operating characteristics curve of the combined BP measurements with finger cuff and arm cuff to detect systolic intra-arterial above 140 mmHg
Discriminative power of the combined BP measurements with finger cuff and arm cuff to detect intra-arterial diastolic hypertension | 30 minutes
  Area under the receiver operating characteristics curve of the combined BP measurements with finger cuff and arm cuff to detect diastolic intra-arterial above 90 mmHg
Accuracy of continuous finger cuff measurements tested against the intra-arterial reference | 30 minutes
  Accuracy of continuous finger cuff BP measurements tested against the intra-arterial reference, according to the ISO standard
Accuracy of intermittent, oscillometric arm cuff BP measurements tested against the intra-arterial reference | 30 minutes
  Accuracy of intermittent, oscillometric arm cuff BP measurements tested against the intra-arterial reference, according to the ISO standard
Accuracy of intermittent, oscillometric calf cuff measurements tested against the intra-arterial reference | 30 minutes
  Accuracy of intermittent, oscillometric calf cuff BP measurements tested against the intra-arterial reference, according to the ISO standard

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire MULLER, Dr, Principal Investigator — CHR Orléans
Locations (3):
- France (3):
  - CHU de NANTES, Nantes
  - CHR Orléans, Orléans
  - CHRU de Tours, Tours

REFERENCES:
- [Derived] Lakhal K, Dauvergne JE, Messet-Charriere H, Nay MA, Kamel T, Muller G, Robert-Edan V, Rozec B, Ehrmann S, Jacquier S, Boulain T. Risk factors for poor performance in finger cuff non-invasive monitoring of arterial pressure: A prospective multicenter study. Anaesth Crit Care Pain Med. 2024 Apr;43(2):101333. doi: 10.1016/j.accpm.2023.101333. Epub 2023 Dec 2. PMID 38048986
- [Derived] Lakhal K, Dauvergne JE, Kamel T, Messet-Charriere H, Jacquier S, Robert-Edan V, Nay MA, Rozec B, Ehrmann S, Muller G, Boulain T. Noninvasive Monitoring of Arterial Pressure: Finger or Lower Leg As Alternatives to the Upper Arm: A Prospective Study in Three ICUs. Crit Care Med. 2023 Oct 1;51(10):1350-1362. doi: 10.1097/CCM.0000000000005945. Epub 2023 May 26. PMID 37232853